CLINICAL TRIAL: NCT02826304
Title: Vaginal Hysterectomy Versus Laparoscopically Assisted Hysterectomy for Large Uteri ( A Pilot Randomized Clinical Trial)
Brief Title: Vaginal Hysterectomy Versus Laparoscopically Assisted Vaginal Hysterectomy for Large Uteri
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Ibrahim Mohamed Ibrahim Ali, lecturer in obstetrics and gynecology, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2016-06-28; First posted 2016-07-07 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Minimally Invasive Hysterectomy in Large Uteri
Keywords: Vaginal Hysterectomy; Laparoscopic assisted vaginal hysterectomy; Large uteri
MeSH Terms: interventions — Hysterectomy, Vaginal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VH (Active Comparator): Vaginal Hysterectomy for uteri larger than 280gm
  Interventions: Procedure: Vaginal hysterectomy
- LAVH (Active Comparator): Laparoscopic assisted vaginal hysterectomy for uteri larger than 280gm
  Interventions: Procedure: Laparoscopic assisted vaginal hysterectomy

INTERVENTIONS:
Procedure: Vaginal hysterectomy — All the cases were performed by the same surgical team
  1. Incision is made at the anterior cervical lip below the bladder reflection
  2. Anterior peritoneal entry .
  3. Douglas pouch entry.
  4. The uterosacral ligaments and the cardinal ligaments are clamped, divided and ligated .
  5. Uterine artery clamping division and ligation
  6. After securing the uterine A., debulking procedures was performed in the form of bisection, coring or myomectomy
  7. Utero-ovarian and round clamping-division and ligation ( in cases where oophorectomy was performed this part was done at the level of the infundibulo-pelvic ligament).
  8. Hemostasis
  9. The vaginal vault is closed after insertion of intraperitoneal drain and
  Arms: VH
Procedure: Laparoscopic assisted vaginal hysterectomy — 1. Uterine manipulator was inserted through the cervix to mobilize the uterus
  2. Veress needle was inserted through the base of the umbilicus
  3. creation of pneumoperitoneum
  4. Insertion of 4 trocars one at the base of umbilicus for the camera and 3 lateral trocars
  5. The round and the utero-ovarian ligament are coagulated and divided.
  6. Dissection through the vesico-uterine space to displace bladder away from the cervix.
  7. Uterine artery was coagulated and divided laparoscopically
  8. anterior colpotomy over the cup of the uterine elevator.
  9. Vaginal part starts with opening of douglas pouch and clamping , division and ligation of uterosacral and cardinal ligaments followed by removal of the uterus and closure of the vault. reinflation to ensure proper hemostasis.
  Arms: LAVH

SUMMARY:
The investigators compare between Vaginal Hysterectomy and Laparoscopically assisted vaginal hysterectomy in cases of large uteri weighing more than 280 gm regarding operative and Postoperative outcomes

DETAILED DESCRIPTION:
Study setting : Ain Shams University Maternity Hospital Study Design : Pilot prospective randomized clinical trial Study population: The patients will be recruited from women presenting to the outpatient clinic of Ain Shams University Maternity Hospital planned to undergo hysterectomy for benign cause according to inclusion/ exclusion criteria which will be mentioned later.

Study duration : the study will be carried out during the period from August 2014 to August 2016.

Sample size: total of 50 cases will be included in the study to be divided into two groups, the first group will undergo vaginal hysterectomy and the second will undergo Laparoscopic assisted vaginal hysterectomy.

intervention: after approval of the ethical committee, a detailed explanation of the procedure will be informed to the participant and after her approval to involve in the study, an informed written consent will be taken. Detailed medical history will be obtained from all participants recruited in the study along with complete clinical examination and necessary laboratory and radiological investigations. Each patient will have a case record form in which the data regarding history, examination, investigations, operation costs and postoperative events will be recorded

ELIGIBILITY:
Inclusion Criteria:

1. Age between 40 and 70 years.
2. Uterine weight more than 280gm. the weight will be estimated sonographically using algebraic formula by Kung and Chang expressed in weights and measurements: weight(g)= 50+(4/3 x π(Pi) x L/2 x W/2 x AP/2) where (L) is the length of the uterus from the dome of the fundus to the level of the external os and (W) is the maximum width of the uterus at the level of the cornua and (AP) is the anteroposterior diameter of the uterus . Both (W) and (AP) will be taken perpendicular to the axis of the uterine length.
3. Presence of a benign cause for hysterectomy. e.g: fibroid uterus, simple endometrial hyperplasia not responding to medical treatment and adenomyosis.

Exclusion Criteria:

1. Patients medically unfit for laparoscopy as severely compromised cardiac patients.
2. Obese patients (BMI>30).
3. Presence of endometriosis.
4. Previous myomectomy
5. Presence of adnexal mass
6. Known or suspected gynecological malignancy.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-08; Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Operative time of the procedure | Range from 90 minutes to 210 minutes
  In case of vaginal hysterectomy, the operative time will be measured from the vaginal incision to closure of the vaginal vault. in cases of Laparoscopic assisted vaginal hysterectomy, the time will be measured from the introduction of the laparoscopic camera port till stitching the laparoscopic incisions after ensuring adequate hemostasis. the time of any concomitant procedures was excluded

SECONDARY OUTCOMES:
Estimated intraoperative blood loss | the operative time of the procedure which range from 90 minutes to 210 minutes
  intraoperative blood loss will be estimated via:
  1. - amount of blood in suction bottle.
  2. - Estimation based on number of soaked gauzes by weighing the gauzes used in the procedure before and after surgery ( each 1mg corresponds to 1ml of blood)
  3. - Drop in postoperative hemoglobin and hematocrit when compared with preoperative values.
Hospital costs | within the period of hospital admission which range from 2 to 8 days
  the costs of the following will be calculated:
  1. - Admission cost which include ward fee, pre and postoperative management costs and extra charges for post surgical complication.
  2. - anesthesia cost which includes expenses of anesthetics during the procedure. C)- operation cost which include operative material fee.
intraoperative complications | the operative time of the procedure which range from 90 minutes to 210 minutes
  1. - need for blood transfusion
  2. - need for laparotomy due to either surgical difficulty or any complication
  3. - Bowel or urinary tract injuries
Postoperative Pain | the first 24hrs after the procedure
  Postoperative pain will be assessed using the visual analogue scale after the procedure by 6hrs, 12hrs and 24hrs.
Postoperative complications | 1 month after the procedure
  1. - Need for blood transfusion
  2. - Vaginal vault or pelvic hematoma
  3. - surgical site infection
  4. - urinary tract infection
  5. - postoperative bowel or urinary tract complications
postoperative hospital stay | range from 24 hours to 168 hours
  the hospital stay will be measured in hours

CONTACTS AND LOCATIONS:
Overall Officials: Fekrya A Salama, PhD, Study Chair — Ain Shams University Maternity Hospital; Ahmed A Tharwat, PhD, Study Director — Ain Shams University Maternity Hospital; Walid E Mohamed, PhD, Study Director — Ain Shams University Maternity Hospital; Ibrahim M Ibrahim, PhD, Study Director — Ain Shams University Maternity Hospital
Locations (1):
- Maternity hospital, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cho HY, Park ST, Kim HB, Kang SW, Park SH. Surgical outcome and cost comparison between total vaginal hysterectomy and laparoscopic hysterectomy for uteri weighing >500 g. J Minim Invasive Gynecol. 2014 Jan-Feb;21(1):115-9. doi: 10.1016/j.jmig.2013.07.013. Epub 2013 Aug 6. PMID 23932973
- [Background] Guvenal T, Ozsoy AZ, Kilcik MA, Yanik A. The availability of vaginal hysterectomy in benign gynecologic diseases: a prospective, non-randomized trial. J Obstet Gynaecol Res. 2010 Aug;36(4):832-7. doi: 10.1111/j.1447-0756.2010.01183.x. PMID 20666953
- [Background] Harb TS, Adam RA. Predicting uterine weight before hysterectomy: ultrasound measurements versus clinical assessment. Am J Obstet Gynecol. 2005 Dec;193(6):2122-5. doi: 10.1016/j.ajog.2005.07.014. PMID 16325627
- [Background] Harmanli OH, Gentzler CK, Byun S, Dandolu MH, Grody T. A comparison of abdominal and vaginal hysterectomy for the large uterus. Int J Gynaecol Obstet. 2004 Oct;87(1):19-23. doi: 10.1016/j.ijgo.2004.06.018. PMID 15464771
- [Background] Hawksley H. Pain assessment using a visual analogue scale. Prof Nurse. 2000 Jun;15(9):593-7. PMID 11129939
- [Background] Johns DA, Carrera B, Jones J, DeLeon F, Vincent R, Safely C. The medical and economic impact of laparoscopically assisted vaginal hysterectomy in a large, metropolitan, not-for-profit hospital. Am J Obstet Gynecol. 1995 Jun;172(6):1709-15; discussion 1715-9. doi: 10.1016/0002-9378(95)91402-1. PMID 7778623
- [Background] Kim HB, Song JE, Kim GH, Cho HY, Lee KY. Comparison of clinical effects between total vaginal hysterectomy and total laparoscopic hysterectomy on large uteruses over 300 grams. J Obstet Gynaecol Res. 2010 Jun;36(3):656-60. doi: 10.1111/j.1447-0756.2010.01185.x. PMID 20598052
- [Background] Lapaire O, Schneider MC, Stotz M, Surbek DV, Holzgreve W, Hoesli IM. Oral misoprostol vs. intravenous oxytocin in reducing blood loss after emergency cesarean delivery. Int J Gynaecol Obstet. 2006 Oct;95(1):2-7. doi: 10.1016/j.ijgo.2006.05.031. Epub 2006 Aug 23. PMID 16934269
- [Background] Nazah I, Robin F, Jais JP, Jeffry L, Lelievre L, Camatte S, Taurelle R, Lecuru F. Comparison between bisection/morcellation and myometrial coring for reducing large uteri during vaginal hysterectomy or laparoscopically assisted vaginal hysterectomy: results of a randomized prospective study. Acta Obstet Gynecol Scand. 2003 Nov;82(11):1037-42. doi: 10.1034/j.1600-0412.2003.00278.x. PMID 14616278
- [Background] Sahin Y. Vaginal hysterectomy and oophorectomy in women with 12-20 weeks' size uterus. Acta Obstet Gynecol Scand. 2007;86(11):1359-69. doi: 10.1080/00016340701657258. PMID 17963064
- [Background] Seracchioli R, Venturoli S, Vianello F, Govoni F, Cantarelli M, Gualerzi B, Colombo FM. Total laparoscopic hysterectomy compared with abdominal hysterectomy in the presence of a large uterus. J Am Assoc Gynecol Laparosc. 2002 Aug;9(3):333-8. doi: 10.1016/s1074-3804(05)60413-6. PMID 12101331
- [Background] Shiota M, Kotani Y, Umemoto M, Tobiume T, Shimaoka M, Hoshiai H. Total abdominal hysterectomy versus laparoscopically-assisted vaginal hysterectomy versus total vaginal hysterectomy. Asian J Endosc Surg. 2011 Nov;4(4):161-5. doi: 10.1111/j.1758-5910.2011.00104.x. Epub 2011 Sep 8. PMID 22776300
- [Background] Teoh TG. Vaginal hysterectomy for the large uterus. Med J Malaysia. 2001 Dec;56(4):460-2. PMID 12014766
- [Background] Wang CJ, Yen CF, Lee CL, Tashi T, Soong YK. Laparoscopically assisted vaginal hysterectomy for large uterus: a comparative study. Eur J Obstet Gynecol Reprod Biol. 2004 Aug 10;115(2):219-23. doi: 10.1016/j.ejogrb.2003.12.021. PMID 15262360
- [Background] Wang CJ, Yuen LT, Yen CF, Lee CL, Soong YK. A simplified method to decrease operative blood loss in laparoscopic-assisted vaginal hysterectomy for the large uterus. J Am Assoc Gynecol Laparosc. 2004 Aug;11(3):370-3. doi: 10.1016/s1074-3804(05)60053-9. PMID 15559351
- [Background] Yen YK, Liu WM, Yuan CC, Ng HT. Comparison of two procedures for laparoscopic-assisted vaginal hysterectomy of large myomatous uteri. J Am Assoc Gynecol Laparosc. 2002 Feb;9(1):63-9. doi: 10.1016/s1074-3804(05)60106-5. PMID 11821608
- [Derived] Mohammed WE, Salama F, Tharwat A, Mohamed I, ElMaraghy A. Vaginal hysterectomy versus laparoscopically assisted vaginal hysterectomy for large uteri between 280 and 700 g: a randomized controlled trial. Arch Gynecol Obstet. 2017 Jul;296(1):77-83. doi: 10.1007/s00404-017-4397-6. Epub 2017 May 15. PMID 28508344